CLINICAL TRIAL: NCT06447337
Title: Examination of a Telemedicine System for Continuous Monitoring of Body Temperature in Adults - a Pilot Study
Brief Title: Continuos Body Temperature Monitoring
Status: Recruiting | Type: Observational
Sponsor: Baby FM Doo (Industry)
Responsible Party: Sponsor
Other Study IDs: BABYFM-010
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Continous body temperature monitoring — The investigational product will be placed on the participants' body in axilar joint and connected to the mobile phone. The values of the current temperature will apear on the monitor and it will be recorded in the database with date and time for each record. In parallel, study staff will occasionally measure the temperature using standard hospital thermometer.

SUMMARY:
This is a nonrandomized, diagnostic, single-center, pilot study, with one group of participants. The aim is to examine the effectiveness and safety of telemedicine system for continuous measurement of body temperature in adults. Up to 40 subjects will participate in this phase of the clinical trial. No stratification, nor randomization of subjects will be performed. Respondents who meet the inclusion criteria will be monitored for up to 72 hours plus 72 hours after removing the device. Namely, the device will be placed on their body and will be there until upt to 72 hours, and then it will be removed. The respondent will be monitored by the team for an additional 72 hours by the person in charge of the examination, for possible side effects.

Sensor will be placed in the axilar joint or a little below on the side. The device will be connected to a mobile phone. Member of the research team (principal researcher/co-researcher/ nurse in charge of examination) measures the temperature of the skin in the opposite armpit manually, ie with a gallium thermometer and records every 30-60 minutes. When body temperature starts to rise, a member of the research team measures the body temperature every 15-30 minutes. After reaching a stable temperature, the temperature is measured every 30-60 minutes. If the subject is given drugs to lower body temperature, the temperature is measured again every 15-30 minutes until the temperature stabilizes to a normal subfebrile state.

ELIGIBILITY:
Inclusion Criteria:

* A person of male or female sex
* Age 18 and over
* Ability to measure the patient's body temperature frequently
* People who are hospitalized due to any type of infection or any other diseases that result in variations in body temperature (rise, fall)
* Completed all potential diagnostics of the hospitalized patient (no interrupting the measurement of the telemedicine device)

Exclusion Criteria:

* Allergic to contact with plastic or silver
* Anatomical anomalies that prevent the placement of the system
* High-risk health conditions, intensive care and the like
* A pacemaker or other device on the skin or implanted in the body that emits light electromagnetic radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 40 eligible participants with disease and/or condition that results in body temperature variation will be included in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between device for continous body temperature monitoring and standard thermometer | up to 72 hours
  The correlation between temperature measurements with the standard hospital thermometer (with galium) is expected to be high

SECONDARY OUTCOMES:
Frequency of device and procedure related adverse events | up to six days
  The number and percentage of adverse events related to the investigational product will be evaluated and summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center of Serbia, Clinic for Infectious and Tropical Diseases, Belgrade, Other/Not Applicable, Serbia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-10-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT06447337/SAP_000.pdf